CLINICAL TRIAL: NCT04997785
Title: A Comparison of Ultrasound-guided Pericapsular Nerve Group (PENG) Block and Parenteral Opioids Alone in Patients With Traumatic Hip Fracture in the Emergency Department: A Multicenter Randomized Controlled Trial
Brief Title: PENG Block for Traumatic Hip Fracture in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, TSAI TOU YUAN, Emergency department physician, Principal Investigator, Dalin Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A10904001
Record Dates: First submitted 2021-07-22; First posted 2021-08-10 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Hip Fractures; Acute Pain; Emergency Department
Keywords: Pericapsular Nerve Group Block (PENG Block)
MeSH Terms: conditions — Hip Fractures; Acute Pain; Emergencies | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided Pericapsular Nerve Group (PENG) Block (Experimental): PENG blocks is performed by Emergency Medicine board-certified emergency physicians (EPs) with standard training program. PENG block is performed using a spinal needle (NIPRO® 21G × 70 mm) at the level of of anterior superior iliac spine, parallel to the inguinal crease, with real-time ultrasound guidance, according to the steps published by Girón-Arango et al in 2018. The investigators use 20 ml of 1% lidocaine for nerve block because this drug has a short onset time, which is adequate to relieve pain before surgical intervention.
  Interventions: Procedure: Ultrasound-guided Pericapsular Nerve Group (PENG) Block
- Intravenous Morphine (Active Comparator): Dosage of intravenous morphine was determined according to 0.1 mg per kg; EPs were instructed to aim to reduce the pain by 50% or per patient request.
  Interventions: Procedure: Ultrasound-guided Pericapsular Nerve Group (PENG) Block

INTERVENTIONS:
Procedure: Ultrasound-guided Pericapsular Nerve Group (PENG) Block — PENG blocks is performed by Emergency Medicine board-certified emergency physicians (EPs) with standard training program. PENG block is performed using a spinal needle (NIPRO® 21G × 70 mm) at the level of of anterior superior iliac spine, parallel to the inguinal crease, with real-time ultrasound guidance, according to the steps published by Girón-Arango et al in 2018. The investigators use 20 ml of 1% lidocaine for nerve block because this drug has a short onset time, which is adequate to relieve pain before surgical intervention.

SUMMARY:
The study is a multicenter single-blinded randomized comparative trial. Adult patients older than 20 years of age presenting with acute hip fracture in emergency department between January 1st, 2021 and December 31st, 2021 will be enrolled. (NOTE: The study was paused temporarily due to local SARS-2 COVID-19 virus pandemic restrictions. Finally, we conducted the study from August 30th, 2021 to May 08th, 2022.) Included patients will receive analgesia with either pericapsular nerve group (PENG) block or intravenous morphine. The primary outcome measure was pain scores (Numeric Rating Scale (NRS) 0 to 10) at rest and with movement. Secondary outcomes were rescue opioids use, complications, length of hospital stay, and patient-reported outcomes.

DETAILED DESCRIPTION:
Study design and setting This is multicenter, randomized controlled comparative trial conducted at Far Eastern Memorial Hospital and Dalin Tzu Chi Hospital, which are academic, level 1 trauma centers in Taiwan. The investigators plan to conduct the study from January 1st to May 8th, 2022. It will be paused temporarily if local coronavirus disease 2019 (COVID-19) virus pandemic restrictions. The trial is registering on ClinicalTrials.gov number. The study was reviewed and approved by the Institutional Review Board. The study conforms to the Consolidated Standards of Reporting Trials (CONSORT) and the CONSORT extension for trials reporting patient- related outcomes.

Selection of participants Patients aged >=20 years presenting to the emergency department (ED) with a diagnosis of traumatic hip fracture from January 1st to May 8th, 2022 will be included. The investigators exclude patients who are aged <20 years, have coagulopathy, injection site infection, allergy to opioids or local anesthetics, initial pulse oximetry measures of oxygen saturation <92%, initial systolic blood pressure < 90 mmHg, chronic opioid use, non-communicative, experiences major trauma, fractures happened > 24 hours, and request conservative(non-operative) treatments. The investigators also exclude patients if the nerve block (NB) providers are unavailable. Written informed consent is acquired from all participants.

Randomization procedures and rationale All the included patients are randomized to either PENG block or intravenous morphine. Because PENG block is a novel technique for regional hip analgesia, well-trained emergency physicians are not available every day. Randomizing patients at the point of ED visit was considered impractical. Therefore, the investigators randomize each visit week before the study begins, and well-trained PENG block providers will be arranged on duty in the weeks randomized for PENG block. The unit of randomization will be the weeks, using random number generation in Microsoft Excel by a statistician who is not involved in the trial.

Study intervention PENG blocks is performed by Emergency Medicine board-certified emergency physicians (EPs) with standard training program. PENG block is performed using a spinal needle (BD® 20G × 90 mm) at the level of of anterior superior iliac spine, parallel to the inguinal crease, with real-time ultrasound guidance, according to the steps published by Girón-Arango et al in 2018. The investigators used 20 ml of 1% lidocaine for nerve block because this drug has a short onset time, which is adequate to relieve pain before surgical intervention. Regimens of regional anesthesia with a longer duration of action are not preferred in our department because delayed onset of regional anesthesia particularly impedes orthopedic assessment in EDs. Dosage of intravenous morphine was determined according to 0.1 mg per kg; EPs were instructed to aim to reduce the pain by 50% or per patient request. They were encouraged to wait for at least 15 minutes after the study procedure before administering additional analgesia.

Outcome measures Primary outcome was postdose NRS pain score at rest and with movement. The NRS for pain with movement was assessed by lifting the affected leg. The examiner assessed NRS score with movement by gently raising the patient's affected limb about 15 degree by flexing the hip with the knee in extension. NRS score was assessed as part of standard care at various timepoints, including at baseline, immediately after the analgesic treatment, at 10, 30, 60, and 120 minutes postdose time points, every 2 h thereafter until discharge from the ED, and at the time of discharge from the ED and arrival at the orthopedic ward before surgery.

Secondary outcomes were postdose quadriceps strength, rescue opiate use, complications, length of ED stay, length of hospital stay, and patient-reported outcomes.

Quadriceps strength was assessed using the knee extension test and Oxford muscle strength scale. Rescue opioid consumption was measured in morphine milligram equivalents (MME) administered over all ED visits during the study timeframe. Any complications or side effects of nerve blocks, including local infection, intravascular injection of local anesthetics and immediate systemic toxicity, will be recorded. In opioid group, any side effects of opioids such as drowsiness, desaturation, nausea and vomiting, delirium, or respiratory distress, will be recorded. Patient-reported outcome defined as patient satisfaction (120 minutes after initial analgesics, patients were asked whether they would choose the same anesthetic handling; "yes" or "no").

Sample size calculation and statistical analyses Sample size could not be calculated, as there is no prior trial on comparison of PENG block and intravenous morphine in patient with hip fractures. This trial will be a pilot trial. Hence, the investigators intend to recruit 200 participants in total using a 1:1 allocation ratio, with 100 participants randomised into each arm. Chi-squared test or Fisher's exact test was used for categorical variables, and Student's t-test was used for continuous variable. Logistic regression was used to analyze data with dichotomous outcomes; p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >20 years presenting to the ED with a diagnosis of traumatic hip fracture during the study timeframe.

Exclusion Criteria:

* are aged <20 years
* coagulopathy
* injection site infection
* allergy to opioids or local anesthetics
* initial pulse oximetry measures of oxygen saturation <92%
* initial systolic blood pressure < 90 mmHg
* chronic opioid use
* non-communicative
* major trauma
* fractures happened > 24 hours
* request conservative(non-operative) treatments.
* The investigators also exclude patients if the NB providers are unavailable.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-05-08 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
Pain intensity difference (PID) | 24 hours
  Pain intensity was investigated at rest and with movement using the 11-point numeric rating-scale (NRS) from 0 (no pain) to 10 (worst pain), and pain-intensity difference(PID) represents the difference in NRS scores between any observation time and the baseline.

SECONDARY OUTCOMES:
postdose quadriceps strength | 24 hours
  Quadriceps strength was assessed using the knee extension test by using Oxford muscle strength scale(from grade 0(no muscle movement) to grade 5(normal strength)) .
Rescue opioid consumption | 24 hours
  measured in morphine milligram equivalents (MME)
Incidence of nerve block complications | 24 hours
  Any complications or side effects of nerve blocks including local infection, intravascular injection of local anesthetics and immediate systemic toxicity.
Incidence of opioid side effects | 24 hours
  Any side effects of opioids such as drowsiness, desaturation, nausea and vomiting, delirium, or respiratory distress.
Patient-reported outcome | 24 hours
  patients were asked whether they would choose the same anesthetic handling; "yes" or "no"

CONTACTS AND LOCATIONS:
Locations (1):
- Dalin Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Chiayi City, Taiwan